CLINICAL TRIAL: NCT00976313
Title: Does Thoracic Epidural Analgesia Influence Urinary Micturition by Patients Undergoing Thoracic Surgery? An Observational, Prospective Study
Brief Title: Does Thoracic Epidural Analgesia Influence Urinary Micturition by Patients Undergoing Thoracic Surgery?
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Dr. Patrick Y. Wuethrich, Universitätsklink für Anästhesiologie und Schmerztherapie, Inselspital, Bern, Switzerland
Other Study IDs: 171/09
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Thoracotomy; Sternotomy
Keywords: thoracic epidural analgesia; urinary micturition; thoracotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: male patients
  Interventions: Procedure: Assessment of urinary micturition after thoracotomy; Other: International Prostate Symptom Score
- 2: female patients
  Interventions: Procedure: Assessment of urinary micturition after thoracotomy; Other: International Prostate Symptom Score

INTERVENTIONS:
Procedure: Assessment of urinary micturition after thoracotomy — Post residual urine volume and voided volume will be assessed with Bladder Scan™ BVI 6100 (Bladder scan, Bothell, WA, USA) will be performed the day before surgery and on day 2 after surgery, with epidural analgesia within segments T2-4 to T10 21,22. Bladder sensitivity will be assessed at strong desire to void. On day 2 the bladder will be filled through the transurethral catheter till the patient signalised a strong desire to void, then the catheter will be removed and spontaneous micturition will be attempted. Voided volume and post void residual will be assessed.
Other: International Prostate Symptom Score — International Prostate Symptom Score (IPSS) for assessment of lower urinary tract symptoms (LUTS) preoperatively

SUMMARY:
Under the influence of epidural analgesia, patients may not feel the urge to urinate, which can result in urinary retention and bladder overdistension.

The use of a transurethral catheter is associated with significant morbidity such as patient discomfort, urinary tract infections, urethral trauma and stricture.

Urodynamic changes under thoracic epidural anaesthesia are still unknown. The aim of this study is to compare lower urinary tract function before and during thoracic epidural analgesia within segments T2 to T10 for postoperative pain treatment in patients undergoing thoracotomy or sternotomy.

DETAILED DESCRIPTION:
Background

1. Background Acute urinary retention is one of the most common complications after surgery and anesthesia. It can occur in patients of both sexes and all age groups and after all types of surgical procedures. It is linked to several factors including increased intravenous fluids, postoperative pain and type of anaesthesia 1.

Micturition depends on coordinated actions between the detrusor muscle and the external urethral sphincter. Motorneurons of both muscles are located in the sacral spinal cord and coordination between them occurs in the pontine tegmentum of the caudal brain stem. Motorneurons innervating the external urethral sphincter are located in the nucleus of Onuf, extending from the S1 to the S3 segment. The detrusor smooth muscle is innervated by parasympathetic fibers, which reside in the sacral intermediolateral cell group and are located in S2-4. Sympathetic fibers innervating the bladder and urethra play an important role in promoting continence and are located in the intermediolateral cell group of the lumbar cord (L1-L4). Most afferent fibers from the bladder enter the sacral cord through the pelvic nerve at segments L4-S2 and the majority are thin myelinated or unmyelinated.

Unlike spinal anesthesia, which is an all or none block, epidural anesthesia has applications ranging from analgesia with minimal motor block to dense anesthesia (differential blockade). Because epidural anesthesia can be performed at various levels of the spinal cord, it is possible to block only a portion of the spinal cord (segmental blockade). Therefore it can be assumed that epidural analgesia within segments Th 4-6 to Th 10-12 has no or minimal influence on the micturition reflex.

There are few studies on the urodynamic effects of various anaesthetic agents 2-8, focused on lumbar epidural anaesthesia. Under the influence of epidural analgesia, patients may not feel the urge to urinate, which can result in urinary retention and bladder overdistension. Overfilling of the bladder can stretch and damage the detrusor muscle.

For example, the use of lumbar epidural analgesia for labor and delivery has frequently been implicated as a causative factor for postpartum urinary retention. This is supported by the fact that these patients demonstrate a difficulty voiding 7. Spinal and epidural opioid administration influence the function of the lower urinary tract by direct spinal action on the sacral nociceptive neurons and autonomic fibres 9.

Long acting local anesthetics administrated intrathecally rapidly block the micturition reflex. Detrusor contraction is restored approximately 7-8 hours after spinal injection of bupivacaine 10. For this reason, bladder catheterisation is a common practice in patients with spinal or epidural anesthesia.

The use of a transurethral catheter is associated with significant morbidity such as patient discomfort, urinary tract infections, urethral trauma and stricture. The risk of infection with a single catheterization is 1-2% and can rise by 3 to 7 % for every additional day with a indwelling catheter 11. Traumatic or prolonged catheterization may lead to urethritis and to urethral strictures 12. There has yet been no consensus for appropriate catheterisation strategy 13-15 during regional anesthesia.

Urodynamic changes under thoracic epidural anaesthesia are still unknown. The aim of this study is to compare lower urinary tract function before and during thoracic epidural analgesia within segments T2 to T10 for postoperative pain treatment in patients undergoing thoracotomy or sternotomy. We expect that a better knowledge on the bladder function under epidural analgesia could lead to a more restrictive use of perioperative transurethral catheters.

Objective

The aim of this study is to compare lower urinary tract function before and during thoracic epidural analgesia within segments T2 to T10 for postoperative pain treatment in patients undergoing thoracotomy or sternotomy. We expect that a better knowledge on the bladder function under epidural analgesia could lead to a more restrictive use of perioperative transurethral catheters.

Hypothesis Thoracic epidural analgesia does not influence urinary micturition in the male and female. Therefore transurethral catheterisation is not mandatory for all patients with thoracic epidural analgesia undergoing thoracic surgery.

Methods

Prospective, open, observational, follow up study. Setting: Department of thoracic surgery, University Hospital Bern

Study population A total of 26 patients (13 men and 13 women per group) undergoing thoracic surgery who receive thoracic epidural anesthesia perioperatively will be needed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Thoracic surgery including thoracotomy and sternotomy
* Thoracic epidural analgesia

Exclusion Criteria

* Contraindications to epidural anesthesia or refusal
* Preoperative residual urine volume > 100ml
* International Prostate Symptom Score (IPSS) > 7
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female patients undergoing thoracotomy or sternotomy
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Differences in postvoid residual urine volume before and during thoracic epidural analgesia | 3 days

SECONDARY OUTCOMES:
Voided volume | 3 days
Maximum bladder capacity | 3 days
Bladder sensitivity (yes/no) at strong desire to void | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wuethrich, MD, Principal Investigator — Dep of Anesthesiologiy and Pain treatment, University Hospital Bern, 3010 Bern, Switzerland
Locations (1):
- Dep of anesthesiology and pain treatment, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Appell RA, England HR, Hussell AR, McGuire EJ. The effects of epidural anesthesia on the urethral closure pressure profile in patients with prostatic enlargement. J Urol. 1980 Sep;124(3):410-1. doi: 10.1016/s0022-5347(17)55474-9. PMID 6159487
- [Background] Kau YC, Lee YH, Li JY, Chen C, Wong SY, Wong TK. Epidural anesthesia does not increase the incidences of urinary retention and hesitancy in micturition after ambulatory hemorrhoidectomy. Acta Anaesthesiol Sin. 2003 Jun;41(2):61-4. PMID 12934418
- [Background] Weiniger CF, Wand S, Nadjari M, Elchalal U, Mankuta D, Ginosar Y, Matot I. Post-void residual volume in labor: a prospective study comparing parturients with and without epidural analgesia. Acta Anaesthesiol Scand. 2006 Nov;50(10):1297-303. doi: 10.1111/j.1399-6576.2006.01122.x. Epub 2006 Sep 15. PMID 16978160
- [Background] Axelsson K, Mollefors K, Olsson JO, Lingardh G, Widman B. Bladder function in spinal anaesthesia. Acta Anaesthesiol Scand. 1985 Apr;29(3):315-21. doi: 10.1111/j.1399-6576.1985.tb02207.x. PMID 3993320
- [Background] Basse L, Werner M, Kehlet H. Is urinary drainage necessary during continuous epidural analgesia after colonic resection? Reg Anesth Pain Med. 2000 Sep-Oct;25(5):498-501. doi: 10.1053/rapm.2000.9537. PMID 11009235
- [Derived] Wuethrich PY, Henning A, Schweizerhof M, Kessler TM, Burkhard FC. Postvoid residuals remain unchanged in patients with postoperative thoracic epidural analgesia after thoracotomy. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):46-50. doi: 10.1097/AAP.0b013e3182030828. PMID 21455089